CLINICAL TRIAL: NCT04438213
Title: Ertugliflozin in Chronic Heart Failure: Cardio-renal and Diuretic Effects
Brief Title: Ertugliflozin in Chronic Heart Failure
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2000027951; MISP59625 (Other Grant/Funding Number: Merck Sharp & Dohme)
Record Dates: First submitted 2020-06-03; First posted 2020-06-18 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Heart Failure
Keywords: Ertugliflozin; Metolazone
MeSH Terms: conditions — Heart Failure | interventions — ertugliflozin; Metolazone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Ertugliflozin (Experimental): Participants will be randomized to six weeks of treatment with either ertugliflozin, metolazone, or a placebo
  Interventions: Drug: Ertugliflozin
- Metolazone (Experimental): Participants will be randomized to six weeks of treatment with either ertugliflozin, metolazone, or a placebo
  Interventions: Drug: Metolazone
- Placebo (Placebo Comparator): Participants will be randomized to six weeks of treatment with either ertugliflozin, metolazone, or a placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ertugliflozin — Participants will be randomized to six weeks of treatment with either ertugliflozin, metolazone, or a placebo
  Arms: Ertugliflozin
Drug: Metolazone — Participants will be randomized to six weeks of treatment with either ertugliflozin, metolazone, or a placebo
  Arms: Metolazone
Drug: Placebo — Participants will be randomized to six weeks of treatment with either ertugliflozin, metolazone, or a placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effects on heart failure signs and symptoms of the use of either ertugliflozin, metolazone or placebo, in conjunction with intravenous loop diuretic use in acute settings and chronic oral loop diuretic therapy.

There are two general purposes for this study. The proposed study is both larger and more rigorous than essentially all PK/PD studies that form the basis of current practice with loop diuretics as well as all studies looking at add-on thiazide therapy (current guideline-recommended adjuvant). The second is to generate a mechanistic understanding of the pleotropic cardio-renal factors with chronic therapy that differentiate ertugliflozin from traditional diuretics particularly in how they maintain reduced blood volume without the complication of over-diuresis and volume depletion.

DETAILED DESCRIPTION:
This is a randomized placebo controlled mechanistic study to understand the utility of ertugliflozin in heart failure patients with or without diabetes, compared to both placebo and the active control metolazone. The broad study design will be designed around evaluation of change in gold standard determined body fluid spaces (blood volume, extracellular fluid, total body water), administering a sodium chloride challenge, and collecting the necessary biospecimens to test our hypotheses. The general study design will randomize to ertugliflozin vs. placebo for a total therapy of 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. A clinical diagnosis of chronic heart failure (either systolic or diastolic)
2. Chronic daily oral loop diuretic dose use
3. eGFR ≥20 mL/min/1.73 m2
4. English speaking participants only
5. Signed informed consent

Exclusion Criteria:

1. Current use or plan to initiate renal replacement therapy or ultrafiltration
2. Significant bladder dysfunction or urinary incontinence
3. Inability to comply with the serial urine collection procedures
4. Current use of a thiazide or thiazide like diuretics or use within 5 half-lives of the drug, including metolazone
5. Current use of a SGLT-2 inhibitor, or in the treating provider's judgement, contraindication to be withdrawn from current use of an SGLT-2 inhibitor
6. Prior heart transplant, critical stenotic valvular disease or complex congenital heart
7. History of type 1 diabetes, diabetic ketoacidosis, "brittle" diabetes or frequent hypoglycemia or severe hypoglycemic episodes requiring emergent intervention (ER visit or EMS response, glucagon administration or forced oral carbs) in the last 3 months
8. History of or current urosepsis or frequent urinary tract infections
9. Anemia with hemoglobin <8g/dL (due to required phlebotomy for the study)
10. Pregnancy or breastfeeding
11. Appears unlikely or unable to participate in the required study procedures, as assessed by the study PI, study coordinator, or designee (ex: clinically-significant psychiatric, addictive, or neurological disease)
12. Inability to give written informed consent or follow study protocol
13. Severe peripheral artery disease, previous amputation, or threatened amputation
14. Life expectancy < 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-03-10 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to day 7 of plasma volume by add-on to loop diuretic therapy | 7 days
  The primary outcome of the chronic effects of add-on placebo, thiazide-like diuretic, or SGLT2 inhibitor is to determine the change in plasma volume from baseline to day 7
Change from baseline to 6 weeks of plasma volume by add-on to loop diuretic therapy | 6 weeks
  The primary outcome of the chronic effects of add-on placebo, thiazide-like diuretic, or SGLT2 inhibitor is to determine the change in plasma volume from baseline to 6 weeks
Natriuretic effect of adjuvant to loop diuretic therapy | 1 day
  The natriuretic effect of each arm with loop diuretic therapy will be measured by the urine sodium output and FeNa.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Testani, MD, Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No